CLINICAL TRIAL: NCT02747147
Title: Multi-Day Evaluation of the TIVA Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Velano Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CP-004
Record Dates: First submitted 2016-04-14; First posted 2016-04-21 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Blood Collections Via Peripheral IV Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A- Control (No Intervention): Group A will have their PIVs assessed daily and record kept of PIV dislodgement or replacement
- B - Device Intervention (Experimental): patients will have their PIVs assessed daily and record kept of PIV displodgement or replacement. patients will additionally have a single blood collection attempted using the study device
  Interventions: Device: TIVA blood collection device

INTERVENTIONS:
Device: TIVA blood collection device — the device is attached to a peripheral IV catheter for use as a direct blood draw device into a vacuum tube or a syringe
  Arms: B - Device Intervention

SUMMARY:
Prospective, randomized, single-center study to evaluate the ability of the device to collect good quality blood samples from patients with peripheral IV access over the length of their stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be admitted to the BWH unit 15 for post-surgical care
* Patient is at least 18 years old
* Patient is willing and physically / cognitively able to sign a written consent form
* Patient is willing and able to complete study questionnaires
* Patient is NOT a prisoner

Exclusion Criteria:

* Active hemodialysis
* Hemolytic disorders (e.g., sickle cell disease)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
% Aspiration reliability | up to 4 days after PIV placement
  blood aspiration with the device is attempted once per day. The % of attempts that are successful will be reported across all attempts
% of Specimen hemolyzed | up to 4 days
  each collected specimen will be analyzed for hemolysis. The hemolysis rate, or % of specimen that are hemolyzed will be reported over all collections.

SECONDARY OUTCOMES:
Avg PIV dwell - hours, mean, range | 1, 2, 3, and 4 calendar days after PIV placement
  note hours between each PIV placement and removal for each patient. compare the the distribution of PIV dwell between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F Mulloy, PhD, RN, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States